CLINICAL TRIAL: NCT00519610
Title: A Study Assessing Patient Outcomes After Placement of H-graft Portacaval Shunts for the Treatment of Portal Hypertension
Brief Title: Assessing Outcome After H-graft Shunt Placement
Acronym: PHTN
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kenneth Luberice, Clinical Research Coordinator, University of South Florida
Other Study IDs: 105982
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Portal Hypertension
Keywords: portal hypertension, H-graft shunt
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: Patients will have charts reviewed for relevant medical information before and after surgery to assess patient outcome after placement of H-graft shunt for the treatment of portal hypertension.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Patients' charts will be reviewed for relevant medical information.

SUMMARY:
The objective of this study is to evaluate the pre-operative symptoms and medical history of patients with portal hypertension who have undergone placement of H-graft portacaval shunts and correlate this with patient outcomes.

DETAILED DESCRIPTION:
Research data will be collected by accessing the Tampa General Hospital medical record charts as well as the Harbourside medical charts, and extracting the necessary research data. The charts will be reviewed for the relevant medical information in order to assess outcomes in patients having H-graft shunts placed for the treatment of portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had H-graft shunts placed for the treatment of portal hypertension.

Exclusion Criteria:

* Patients under the age of 18 will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with portal hypertension
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-07; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to evaluate the pre-operative symptoms and medical history of patients with portal hypertension who have undergone placement of H-graft portacaval shunts and correlate this with patient outcomes. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Rosemurgy, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital/University of South Florida, Tampa, Florida, United States